CLINICAL TRIAL: NCT01017289
Title: A Study Evaluating the Quantum - Composite Nailing System for Intramedullary Fixation of Humerus Fractures
Brief Title: Intramedullary Fixation of Humerus Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: N.M.B. Medical Applications Ltd (Industry)
Responsible Party: Michael Bernstein, Senior Orthopedic Surgeon, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N.M.B. P Q REV I 03.09
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Humeral Fractures; Pathological Fractures
MeSH Terms: conditions — Humeral Fractures; Fractures, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quantum (Experimental): In this single arm study, the Quantum nailing system will be used in all patients.
  Interventions: Device: Quantum

INTERVENTIONS:
Device: Quantum — Treatment of humerus fracture (according to the mentioned indications) with the Quantum Intramedullary Nailing System.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the composite Nail - the Quantum interlocking intramedullary nailing system in the reduction of humeral fractures.

DETAILED DESCRIPTION:
The study will include 20 patients who have an acute mid shaft diaphyseal humeral fracture due to injury. The patients will undergo lateral and AP X- ray evaluation of the fracture. Following General anesthesia, closed reduction of the fracture will be performed. It will be followed by nail insertion, percutaneously, according to standard surgical techniques, with the help of the insertion handle. Following insertion the nail will be locked both distally and proximally using interlocking screws. The nail and screws insertion will be monitored by fluoroscopy. Patients will remain under follow up for 6 months following the procedure. In the follow up sessions the fracture will be evaluated by fluoroscopy or X-ray for correct bone alignment, callus formation, and fracture union.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.
* Mid shaft diaphyseal fracture
* Acute fracture

Exclusion Criteria:

* Patients with metabolic or hormonal diseases that could affect bone healing such as diabetes.
* Ongoing infection in fracture site.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Bone union and callus formation | up to 6 months
Bone alignment | up to 6 months
Nail and screws resistance over time | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berenstein, md, Principal Investigator — Rabin hospital
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel